CLINICAL TRIAL: NCT01122472
Title: Double Blind Randomized Phase III Study of Lenalidomide Maintenance Versus Placebo in Responding Elderly Patients With DLBCL and Treated With R-CHOP in First Line
Brief Title: Study of Lenalidomide Maintenance Versus Placebo in Responding Elderly Patients With DLBCL and Treated With R-CHOP
Acronym: REMARC
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: The Lymphoma Academic Research Organisation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: REMARC
Record Dates: First submitted 2010-04-08; First posted 2010-05-13 (Estimated); Last update posted 2021-07-26 (Actual); Status verified 2021-07

CONDITIONS: Lymphoma; Diffuse Large B-cell Lymphoma
Keywords: lenalidomide (Revlimid); diffuse large B-cell lymphoma; phase III study; after R-CHOP; Maintenance treatment; Maintenance
MeSH Terms: conditions — Lymphoma; Lymphoma, Large B-Cell, Diffuse | interventions — Lenalidomide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lenalidomide (Experimental): Lenalidomide daily for 3 weeks every 4 weeks for 24 months
  Interventions: Drug: Lenalidomide
- Placebo (Placebo Comparator): Placebo daily for 3 weeks every 4 weeks for 24 months
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Lenalidomide — Daily for 3 weeks every 4 weeks for 24 months
  Other Names: Revlimid
  Arms: Lenalidomide
Drug: Placebo — Daily for 3 weeks every 4 weeks for 24 months
  Arms: Placebo

SUMMARY:
This study is designed as a phase III, randomized, double-blind, placebo-controlled trial to explore the effect of maintenance therapy with lenalidomide versus placebo on progression-free survival (PFS) in patients treated with R-CHOP responding to induction therapy

For the primary efficacy variable, PFS, an improvement in median PFS from 38.6 months for Treatment Arm B to 54 months for Treatment Arm A (corresponding to a 2-year PFS of 65% vs 73.6%), is considered clinically relevant.

DETAILED DESCRIPTION:
Patients should have received at least 6 and up to 8 cycles of the R-CHOP 14 or R-CHOP 21 regimen or 6 R-CHOP-14 or -21 completed by 2 Rituximab alone in accordance to local preferences.

Patients can be registered to participate in the study at two time points:

* At time of initial diagnosis and study enrolment (signature of informed consent) before the first cycle of treatment with R-CHOP.
* At randomization (signature of informed consent) after treatment in first line with R-CHOP and have reached at least PR or CR.

Evaluation of the response to R-CHOP must be in accordance with Revised Response Criteria for Malignant Lymphoma(2007).

Stratification: Before randomization, the patients will be stratified according to the country and the response to R-CHOP (PR vs CR).

Randomization: Patients in CR/PR after R-CHOP will be randomized to maintenance therapy with lenalidomide or placebo.

ELIGIBILITY:
Ages Eligible for Study: Between 60 and 80 years old

Genders Eligible for Study: Both

Accepts Healthy Volunteers: No

Inclusion Criteria:

For patients registered at the time of initial diagnosis

* Patient with histologically proven CD20+ diffuse large B cel LYMPHOMA (DLBCL) 5WHO classification 2008) including clinical subtypes (primitive mediastinal, intravascular, etc.). Patients with De Novo Transformed DLBCL from low grade lymphoma (Follicular, other..) may also be included. Patients with DLBCL associated with some small cell infiltration in bone marrow may also be included Or CD20+ B-cell lymphoma with intermediate features between DLBCL and Burkitt or with intermediate features between DLBCL and classical Hodgkin lymphoma Or CD20+ Follicular lymphoma grade 3B Or CD20+ Aggressive B-cell lymphoma unclassifiable
* previous untreated with chemo- or radiotherapy

For patients registered after response evaluation to first line treatment with R-CHOP:

* Patient with histologically proven CD20+ diffuse large B cell LYMPHOMA (DLBCL) 5WHO classification 2008) including clinical subtypes (primitive mediastinal, intravascular, etc.). Patients with De Novo Transformed DLBCL from low grade lymphoma (Follicular, other..) may also be included. Patients with DLBCL associated with some small cell infiltration in bone marrow may also be included Or CD20+ B-cell lymphoma with intermediate features between DLBCL and Burkitt or with intermediate features between DLBCL and classical Hodgkin lymphoma Or CD20+ Follicular lymphoma grade 3B Or CD20+ Aggressive B-cell lymphoma unclassifiable
* Have reached a CR or PR after first line treatment with at least 6 cycles of R-CHOP 14 regimens and up to 8 cycles of R-CHOP21
* Previously untreated with Radiotherapy

For all patients:

* aged from 60 to 80 years at time of registration
* Ann Arbor stages II-IV at time of initial diagnosis
* aaIPI> 1 at time of initial diagnosis
* ECOG performance status 0-2
* Minimum life expectancy of 3 months
* Following laboratory values at screening:

  * ANC≥ 1000.10^6/L and Platelets≥60000.10^6/L
  * AST<5*ULN, ALT<5*ULN, Total Bilirubin<1,5*ULN
  * Creatinine clearance>30mL/min
* Women are are using effective contraception, are not pregnant and agree not to become pregnant during participation in the trial and after end of study. Men agree not to father a child during participation in the trial and during the 12 months thereafter.
* Having previously signed a written informed consent form

Exclusion Criteria:

* Any other histological type of Lymphoma, Burkitt included.
* Any history of treated or non treated small B-cell lymphoma
* Central nervous system or meningeal involvement by lymphoma
* Contraindication to any drug contained in the chemotherapy regimen Myocardial infarction during last 3 months or unstable coronary disease or uncontrolled chronic symptomatic congestive heart insufficiency NYHA III-IV
* Uncontrolled hypertension
* Uncontrolled diabetes mellitus as defined by the investigator
* Active systemic infection requiring treatment
* previously known HIV positive serology
* Active hepatitis B or C
* Prior history of malignancies other than lymphoma within 3 years
* Serious medical or psychiatric illness

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 650 (Actual)
Dates: Start 2009-04; Primary Completion 2016-06 (Actual); Study Completion 2019-09 (Actual)

PRIMARY OUTCOMES:
Progression-Free-Survival (PFS) | Final PFS analysis will be realized when the number of events (160) has been reached or at the latest when the last patient into the study will finish follow up. The approximate schedule will be 75 months after the first patient randomized.
  PFS will be measured from the date of randomization to the date of first documented disease progression or death. Progression data will be assigned to the earliest time when any progression is observed without prior missing assessments during the study up to the end of the follow up phase.

SECONDARY OUTCOMES:
Overall survival (OS) | 5 years
  From the date of randomization to the date of death from any cause Interim analysis of OS will be performed at the time of the PFS final analysis; it is projected to have 97 deaths at this time. Final analysis of OS at the end of the study, defined by the last visit of follow-up for the last patient randomized, 5 years after its randomization
Event-Free Survival (EFS) | 5 years
  From the date of randomization to the date of first documented disease progression, relapse, initiation of new anti-lymphoma therapy or death from any cause Interim analysis of EFS will be performed at the time of the PFS final analysis. Final analysis of OS at the end of the study, defined by the last visit of follow-up for the last patient randomized, 5 years after its randomization
Response rate at the end of maintenance treatment | 24 months
Percentage of patients who convert from PR (partial response) to CR (complete response) | 24 months
Safety of lenalidomide in maintenance | 5 years
  Toxicities occured during maintenance phase will be measured and reported from grade 2 for infection and neurological toxicities and from grade 3 for other toxicities according to CTCAE v3
PFS2 | 5 years
  From randomization to objective tumor progression on next-line treatment or death from any cause

CONTACTS AND LOCATIONS:
Locations (157):
- Australia (15):
  - Bendigo Hospital, Bendigo
  - Concord Repatriation General Hospital, Concord
  - Flinders Medical Centre - Repatriation General Hospital, Daw Park
  - St Vincent's Hospital, Melbourne, Fitzroy
  - Frankston Hospital Monash Medical Centre, Frankston
  - Fremantle Hospital, Fremantle
  - Canberra Hospital, Garran
  - Austin Hospital, Heidelberg
  - Royal Hobart Hospital, Hobart
  - Mater Misericordiae Hospital - Calvary Mater NewCastle, Hunter
  - St George Hospital, Kogarah
  - Sir Charles Gardiner Hospital, Nedlands
  - Gold Coast Hospital, Southport
  - Albury Base Hospital/Murray Valley Private Hospital, Wodonga
  - Queen Elizabeth Hospital, Woodville
- Austria (10):
  - LKH Feldkirch, Feldkirch
  - Medizinische Universität Innsbruck für Innere Medizin, Innsbruck
  - LKH Leoben-Eisenerz Department für Hämato-Onkologie, Leoben
  - Krankenhaus Barmherzigen Schwestern Linz - Abteilung für Inner, Linz
  - Krankenhaus der Elisabethinen Linz GmbH, Linz
  - AKh Linz - Innere Medizin 3 - Zentrum für Hämatologie un, Linz
  - Universitätklinik der PMU Salzburg - Für Innere Medizin III, Salzburg
  - Landeskrankenhaus Steyr - Innere Medizin II, Steyr
  - Uniersitätsklinik f. Innere Medizin I, Vienna
  - Klinikum Wels-Grieskirchen GmbH, Wels
- Belgium (26):
  - ZNA Middelheim, Antwerp
  - ZNA Stuivenberg, Antwerp
  - Hopital Saint Joseph, Arlon
  - A.Z. Sint Jan AV, Bruges
  - CHU Brugmann, Brussels
  - Institut Jules BORDET, Brussels
  - Universite Catholique de Louvain Saint Luc, Brussels
  - CH Notre Dame, Charleroi
  - CHU Charleroi-Vesale, Charleroi
  - Centre de Sante des Fagnes, Chimay
  - Universitair Ziekenhuis Gent, Ghent
  - Clinique Notre Dame de Grace, Gosselies
  - Hopital Jolimont, Haine-Saint-Paul
  - CH Hutois, Huy
  - AZ VUB, Jette
  - AZ Groeninge - Campus Maria s Voorzienigheid, Kortrijk
  - CHR de la Citadelle, Liège
  - CHU de Liege, Liège
  - CHU Ambroise Pare, Mons
  - Clinique Saint Joseph, Mons
  - Hopital Sainte Elisabeth, Namur
  - Clinique Saint Pierre, Ottignies
  - Heilig Hart Ziekenhuis, Roeselare
  - CH de la Tourelle-Peltzer, Verviers
  - A.Z. Sint-Augustinus, Wilrijk
  - Universite Catholique de Louvain Mont Godinne, Yvoir
- France (73):
  - CHR de la Région d'Annecy, Annecy
  - CH Antibes-Juan les Pins, Antibes
  - CH d'Arras, Arras
  - Hopital Henri DUFFAUT, Avignon
  - Hopital de BAYONNE, Bayonne
  - CHG Mail Pierre Charlot, Blois
  - Hôpital d'Avicenne, Bobigny
  - Hopital Jean VERDIER, Bondy
  - Polyclinique Bordeaux Nord Aquitaine, Bordeaux
  - Hopital DUCHENNE, Boulogne-sur-Mer
  - CH de Bourg-en-Bresse, Bourg-en-Bresse
  - Centre Hospitalier de Brive, Brive-la-Gaillarde
  - Centre François Baclesse, Caen
  - CHU Clémenceau- Côte de Nacre, Caen
  - CH de Cannes, Cannes
  - Hôpital de Châlon, Chalon-sur-Saône
  - Centre Hospitalier, Chambéry
  - CH Chartres, Chartres
  - Hopital Antoine Béclère, Clamart
  - Hôpital des instructions des Armées PERCY, Clamart
  - Hopital Louis Pasteur, Colmar
  - CH de Compiègne, Compiègne
  - Hopital Sud Francilien, Corbeil-Essonnes
  - CH Henri Mondor, Créteil
  - CHU le Bocage, Dijon
  - CH de Dunkerque, Dunkirk
  - CHI Evreux, Évreux
  - CHI Fréjus Saint Raphaêl, Fréjus
  - Institut Daniel Hollard, Grenoble
  - Centre Hospitalier de Guéret, Guéret
  - CHG La Rochelle, La Rochelle
  - Hopital André Mignot, Le Chesnay
  - Hopital Bicêtre, Le Kremlin-Bicêtre
  - Clinique Victor Hugo - Centre Jean Bernard, Le Mans
  - CHU de Lens, Lens
  - Hôpital Saint Vincent de Paul, Lille
  - CHRU de Lille, Lille
  - Hopital DUPUYTREN, Limoges
  - Clinique de la Sauvegarde, Lyon
  - Centre Léon Bérard, Lyon
  - Institut Paoli Calmettes, Marseille
  - Hopital Nord, Marseille
  - CH les CHANAUX, Mâcon
  - CHG Meaux, Meaux
  - CH Marc JACQUET, Melun
  - Hopital Notre Dame de Bon Secours, Metz
  - CRLC Val d'Aurelle, Montpellier
  - Centre Azuréen de Cancérologie, Mougins
  - Hopital Emile Muller- CHU Mulhouse, Mulhouse
  - Hôpital Américain de Paris, Neuilly-sur-Seine
  - Centre Antoine Lacassagne, Nice
  - CHU de Nice, Nice
  - Hopital Saint Antoine, Paris
  - Hôtel Dieu, Paris
  - Institut Curie, Paris
  - Hopital St-Louis, Paris
  - Hopital de la Pitié Salpetrière, Paris
  - Hopital NECKER, Paris
  - CH de Perpignan, Perpignan
  - Centre Hospitalier Lyon Sud, Pierre-Bénite
  - CH René DUBOS, Pontoise
  - Hopital Robert DEBRE, Reims
  - Centre Henri BECQUEREL, Rouen
  - Clinique Mathilde, Rouen
  - Centre René Huguenin, Saint-Cloud
  - CHG Saint Germain, Saint-Germain-en-Laye
  - CHI Toulon La Seyne-sur-mer, Toulon
  - CHU Purpan Pav. Dieulafoy, Toulouse
  - Hopital de Troyes, Troyes
  - CH Valence, Valence
  - CH de Valenciennes, Valenciennes
  - CHU Nancy Brabois, Vandœuvre-lès-Nancy
  - Institut Gustave ROUSSY, Villejuif
- Israel (7):
  - Haemek Medical Center, Afula
  - Barzilai Medical Center, Ashkelon
  - Soroka, Beersheba
  - Bnai-Zion medical center, Haifa
  - Meir Medical Center, Kfar Saba
  - Rabin Medical Center - Beilinson Hospital, Petah Tikva
  - Kaplan Medical Center, Rehovot
- Poland (5):
  - SPZOZ Zespol Szpitali Miejskich w Chorzowie, Chorzów
  - Klinika Hematologii Collegium Medicum UJ, Krakow
  - Oddzial Chorob Rozrostowych Regionalny Osrodek Onkologiczny, Lodz
  - Medical University of Warsaw, Warsaw
  - Klinika Nowotworow Ukladu Chlonnego- Centrum Onkologii, Warsaw
- Portugal (4):
  - Hospitais da Universidade de Coimbra, Coimbra
  - Instituto Português de Oncologia de Lisboa de Francisco Gentil, Lisbon
  - Hospital de Santa Maria, Lisbon
  - IPO - Francisco Gentil - Porto, Porto
- Spain (16):
  - Complejo Hospitalario Universitario de A Coruna, A Coruña
  - Hospital Universitario Fundacion Alcorcon, Alcorcón
  - Hospital Clinic Barcelona, Barcelona
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hopital Universitario Virgen de la Arrixaca, El Palmar
  - Hopital de Jerez (S.A.S), Jerez de la Frontera
  - Hospital de Leon, León
  - Hospital 12 de Octubre, Madrid
  - Hospital Général Universitario Gregorio Maranon, Madrid
  - Hospital Universitario - La Paz, Madrid
  - Hospital Morales Meseguer, Murcia
  - Hospital Central Asturias, Oviedo
  - Hospital Clinico Salamanca, Salamanca
  - Universitario Marques de Valdecilla, Santander
  - Hospital Joan XXIII, Tarragona
  - Hospital Mutua de Terrassa, Terrassa
- Centre Hospitalier Universitaire Vaudois, Lausanne, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Montagne A, Bertho G, Papastergiou T, Chartier L, Ricci R, Jardin F, Ghesquieres H, Rossi C, Morschhauser F, Haioun C, Ribrag V, Feugier P, Brisou G, Oberic L, Gaulard P, Giraud N, Bennani Y, Thieblemont C, Baud V. Risk stratification of patients with diffuse large B-cell lymphoma using plasma NMR-based metabolomics at diagnosis. Blood Adv. 2026 Jan 27;10(2):358-366. doi: 10.1182/bloodadvances.2025017248. PMID 41056515
- [Derived] Beldi-Ferchiou A, Jais JP, Ghesquieres H, Casasnovas RO, Tilly H, Fruchart C, Morschhauser F, Haioun C, Lazarovici J, Perrot A, Nicolas-Virelizier E, Salles G, Godard N, Zamali I, De Colella JS, Claudel A, Corront B, Oberic L, Briere J, Gaulard P, Thieblemont C, Delfau-Larue MH. Lenalidomide maintenance fails to overcome the unfavourable prognosis of low NK-cell counts in rituximab-chemotherapy responsive elderly DLBCL patients: A LYSA group study. Br J Haematol. 2023 Apr;201(2):256-266. doi: 10.1111/bjh.18642. Epub 2023 Feb 6. PMID 36740991
- [Derived] Girum KB, Rebaud L, Cottereau AS, Meignan M, Clerc J, Vercellino L, Casasnovas O, Morschhauser F, Thieblemont C, Buvat I. 18F-FDG PET Maximum-Intensity Projections and Artificial Intelligence: A Win-Win Combination to Easily Measure Prognostic Biomarkers in DLBCL Patients. J Nucl Med. 2022 Dec;63(12):1925-1932. doi: 10.2967/jnumed.121.263501. Epub 2022 Jun 16. PMID 35710733
- [Derived] Cottereau AS, Meignan M, Nioche C, Capobianco N, Clerc J, Chartier L, Vercellino L, Casasnovas O, Thieblemont C, Buvat I. Risk stratification in diffuse large B-cell lymphoma using lesion dissemination and metabolic tumor burden calculated from baseline PET/CTdagger. Ann Oncol. 2021 Mar;32(3):404-411. doi: 10.1016/j.annonc.2020.11.019. Epub 2020 Dec 3. PMID 33278600
- [Derived] Vercellino L, Cottereau AS, Casasnovas O, Tilly H, Feugier P, Chartier L, Fruchart C, Roulin L, Oberic L, Pica GM, Ribrag V, Abraham J, Simon M, Gonzalez H, Bouabdallah R, Fitoussi O, Sebban C, Lopez-Guillermo A, Sanhes L, Morschhauser F, Trotman J, Corront B, Choufi B, Snauwaert S, Godmer P, Briere J, Salles G, Gaulard P, Meignan M, Thieblemont C. High total metabolic tumor volume at baseline predicts survival independent of response to therapy. Blood. 2020 Apr 16;135(16):1396-1405. doi: 10.1182/blood.2019003526. PMID 31978225
- See also: Related Info — http://www.lysa-lymphoma.org/